CLINICAL TRIAL: NCT03714295
Title: Impact of Interdental Brushing on the Evolution of Supra-gingival Bacterial Flora in Healthy Subjects Aged 18 to 35 Years (BACTERIB)
Brief Title: Impact of Interdental Brushing on the Evolution of Supra-gingival Bacterial Flora (BACTERIB)
Acronym: BACTERIB
Status: Completed | Type: Observational
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Denis Bourgeois, Sponsor, Claude Bernard University
Other Study IDs: BACTERIB
Record Dates: First submitted 2018-10-15; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Use of interdental brushes: The group use interdental brushes one time each day and wash teeth with a classical brush two times a day
  Interventions: Other: Use of interdental brushes
- No use of interdental brushes: The group wash teeth with a classical brush two times a day
  Interventions: Other: Use of interdental brushes

INTERVENTIONS:
Other: Use of interdental brushes — No intervention they just use interdental brushes as it should be done routinely

SUMMARY:
In France, two-thirds of adults over 35 years of age have at least a periodontal disease. The etiology is the accumulation of dental plaque, especially in interdental spaces. The cleaning of interdental spaces is particularly complex. This accumulation of dental plaque is at the origin of a modification of the bacterial flora in favor of periodontopathogenic bacteria. These pathogens can induce within the periodontal tissues an immune and inflammatory reaction that cause tissue degradation. The majority of studies focus on people over 30 years of age with gingivitis or periodontitis. However, young adults, in whom the initial or even reversible stages of periodontal disease are the most frequent, should be the preferred target of preventive measures for this pathology.

The main objective of this study is to quantify, in healthy patients, the evolution of the supragingival bacterial flora, in the interdental spaces, following the daily passage of brushes with the adapted diameter and single passage. The secondary objective is to evaluate the qualitative change in the bacterial flora (proportions of periodontal bacteria / commensal bacteria) following the interdental cleaning.

ELIGIBILITY:
Inclusion Criteria:

* having teeth at the 4 interdental sites studied (15-16, 25-26, 35-36, 45-46),
* reporting a minimum of two daily toothbrushes,
* having a good understanding of the French language,
* accepting the terms of the study and signing written informed consent,
* in good general health (opinion of the investigator) without significant clinical abnormality and medical history.

Exclusion Criteria:

* Smoking patients (daily consumption greater than or equal to 1 cigarette),
* patients with pathologies: diabetic, haemophilia, anticoagulant, platelet antiaggregant, pregnant and lactating women,
* patients with a history of periodontal treatments,
* patients with mandibular fixed orthodontic appliances and or maxillary, masticatory coefficient less than 80%,
* patients who have taken antibiotics in the past 3 months,
* patients using interdental brushes on a regular basis (more than once a week) in addition to brushing teeth or mouthwash ,
* patients at risk for infectious endocarditis,
* patients unable to answer questions,
* non-cooperative patients,
* patients requiring geographic mobility compromising evaluation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: - Subjects aged from 18 to 35 years in good health
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Enumeration of periodontal pathogens in interdental microbiota | 3 months
  Quantitative RT-PCR analyses for A. viscosus, S.mitis, Streptococcus sp., V. parvula, A. odontolyticus, E. corrodens, C. sputigena, C. ochracea, C. concisus, A. actino a, A. actino b, S. sobrinus.- et des bactéries pardonthopathogènes - C. gracilis, C. rectus, P. intermedia, P. nigrescens, P. micros, F. nuc, P. gingivalis, T. forsythensis, T. denticola, S. mutans, and Lactobacillus spp. in the interdental microbiota.

SECONDARY OUTCOMES:
Enumeration of periodontal pathogens in interdental microbiota of young adults using or not interdental brushes by real-time PCR | 3 months
  Quantitative RT-PCR analyses for A. viscosus, S.mitis, Streptococcus sp., V. parvula, A. odontolyticus, E. corrodens, C. sputigena, C. ochracea, C. concisus, A. actino a, A. actino b, S. sobrinus.- et des bactéries pardonthopathogènes - C. gracilis, C. rectus, P. intermedia, P. nigrescens, P. micros, F. nuc, P. gingivalis, T. forsythensis, T. denticola, S. mutans, and Lactobacillus spp. in the interdental microbiota of young adults using or not interdental brushes.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Bourgeois, Pr, Study Director — University Lyon
Locations (1):
- University Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No